CLINICAL TRIAL: NCT03670485
Title: A Prospective Study of Compensatory Medical Device Pivotal Clinical Study to Assess the Safety and Efficacy of the 4 Channel NMES, Multicenter Study
Brief Title: To Assess the Safety and Efficacy of the 4 Channel NMES Compensatory Medical Device in Swallowing, Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1806-475-001
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Dysphagia
Keywords: stroke; cervical spinal cord injury
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revised sequential activation protocol (Experimental): Apply 4 channel electrical stimulation device with a revised sequential activation protocol.
  It sequentially activates Rt. suprahyoid m (ch 1), Lt. suprahyoid m (ch 2), thyrohyoid m (ch 3), sternothyroid m (ch 4) with 4 channel electrical stimulation device.
  Interventions: Device: 4 channel Electrical Stimulation Device
- control subject (No Intervention): Apply 4 channel electrical stimulation device without any stimulation

INTERVENTIONS:
Device: 4 channel Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition
  Arms: Revised sequential activation protocol

SUMMARY:
This study is a confirmation study to prepare clinical trials to evaluate the safety and effectiveness of 4-channel electric stimulation therapy devices as a newly developed function for the treatment of dysphagia disorders. The purpose of this study is to validate the 4ch NMES device.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of patient group: who has a dysphagia symptom and confirmed by video-fluoroscopic swallowing study
* Intervention: applied electrical stimulation by a "Synchronized Electrical Stimulation Device(SESD)"
* Main outcome measures: videofluoroscopic parameters, EQ-5D (EuroQoL-5D) questionnaire, II. M. D Anderson dysphagia inventory

ELIGIBILITY:
Inclusion Criteria:

* patient who do not belong to the criteria excluded for subjects aged 19 years or older
* Patient who is confirmed to be dysphagia by videofluoroscopy
* Patients who need clinical application of electrical stimulation therapy equipment for dysphagia. ex) stroke, cervical spinal cord injury
* Those voluntarily agreeing to the clinical trial

Exclusion Criteria:

* Patient who refuse inspection, do not agree
* Simple "Commend obey", first step is impossible
* When instructions can not be executed due to dementia, psychiatric disorders, etc.
* Dysphagia occurs due to respiratory failure, neck surgery, etc.,
* Pregnant women and lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
The Modified Barium Swallow Impairment Profile (MBSImP™©) | Change from Baseline without stimulation at within 1 weeks with electrical stimulation applied
  total score 0 from 55, 55 is worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Bundang, South Korea

IPD SHARING:
Plan to Share IPD: No